CLINICAL TRIAL: NCT05074654
Title: Reliability and Validity of Urdu Version of Neck Pain and Disability Scale (NPAD)
Brief Title: Urdu Version of Neck Pain and Disability Scale (NPAD)
Status: Completed | Type: Observational
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Other Study IDs: REC-FSD-00243
Record Dates: First submitted 2021-09-29; First posted 2021-10-12 (Actual); Last update posted 2022-01-19 (Actual); Status verified 2022-01

CONDITIONS: Neck Pain; Neck Disorder
Keywords: Neck pain and disability scale; Pain; Disability; Reliability and validity; population with neck pain
MeSH Terms: conditions — Neck Pain; Pain

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In this study, the examiners will investigate the reliability and validity of neck pain and disability scale in Urdu language in Pakistani patients with neck pain and related disability.

DETAILED DESCRIPTION:
This study's objective is to translate the Neck Pain and Disability Scale (NPAD) into Urdu and evaluate its reliability and validity in Pakistani neck pain individuals. This cross-sectional survey will employ convenience sampling to choose participants.

This study's findings will assist determine the NPAD's reliability and validity in individuals with neck pain and impairment. This scale's reliability will be evaluated utilising internal consistency and test-retest methods. Cronbach's alpha value checks internal consistency. The interclass correlation will be used to examine the test-retest reliability.

ELIGIBILITY:
Inclusion Criteria

* Individuals including both male and females between age 18 and 65 years.
* Participants with non-specific chronic pain of neck (>3 months in duration).
* Individuals with sufficient knowledge and understanding of Urdu language.

Exclusion Criteria

* Individuals with history of cervical surgery.
* Individuals with cervical myelopathy or radiculopathy, regional tumors, disc herniation, vertebral fractures, traumatic injuries, cardiovascular and pulmonary diseases, pregnancy or any behavioral problems were excluded
* Individuals with any pertinent comorbidities including heart attack, cancer, cognitive impairment or infection were also excluded. herniation, vertebral fractures, traumatic injuries, cardiovascular and pulmonary diseases, pregnancy or any behavioral problems were excluded
* Individuals with any pertinent comorbidities including heart attack, cancer, cognitive impairment or infection were also excluded.

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: People with non-specific chronic neck pain that interferes with their social, recreational, functional, vocational and emotional aspects of living. Chronic non-specific neck pain is related to limited cervical mobility, impaired function, neck muscles myofascial pain syndrome, and stress at work. The aforementioned factors are strongly related and may lead to a negative impact on health-related quality of life.
Sampling Method: Non-Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-10-15 (Actual); Study Completion 2021-10-15 (Actual)

PRIMARY OUTCOMES:
Neck Pain and Disability scale | 1st day
  The Neck Pain and Disability Scale is a multidimensional configuration measure that contains a 20-item questionnaire to assess neck pain and disability. This scale measures neck mobility and severity difficulties, as well as the impact of neck injuries on everyday activities.

SECONDARY OUTCOMES:
Neck Disability Index | 1st day
  This tool assesses the quality of pain, lifting, personal care, job activities, headaches, sleep, drive, and leisure activities. Each item is graded from 0 to 5. The Neck Disability Index is a one-dimensional evaluation instrument designed to show how neck pain affects activities and capability. This is a reliable and useful self-declared estimate tool for neck problems. This scale may be used to assess a patient's current condition and progress throughout therapy.
Pain Disability Index | 1st day
  The Pain Disability Index is an authentic simple measure of indiscriminate pain and disability and is used for the evaluation of the influence of pain on the capability of an individual's participation skills in everyday important activities. It has also been used in assessment of the patients before interventions and then monitoring them over time to evaluate the efficacy of interventions. This scale comprises of 7 sections which include family, home responsibilities, recreation, occupation, sexual and social activities, self-care and life support and these items are totaled into a score between 0-70.
Visual Analogue Scale | 1st day
  The Visual Analogue Scale is a unique instrument for assessing chronic and acute pain as well as pain perception. It is a scale that assesses the frequency and severity of pain experienced by a person. Patient selects a position on the line that best represents their pain perception.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Kashif, Study Chair — Riphah International University
Locations (1):
- Ripah International University, Faisalabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No